CLINICAL TRIAL: NCT06261983
Title: Diagnostic Value of Sentinel Node Biopsy Guided by Magnetic Probe in Squamous Cell Oral Carcinoma: a Prospective Observational Study
Brief Title: Magnetic Localization of Sentinel Nodes in Squamous Cell Oral Carcinoma.
Acronym: SentiMag
Status: Recruiting | Type: Observational
Sponsor: Hospital Donostia (Other)
Responsible Party: Principal Investigator, Josue Hernando, PhD, DDS, Hospital Donostia
Other Study IDs: 2019111032
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Diagnostic Value of Sentinel Node Biopsy Guided by Magnetic Probe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosed with oral squamous cell carcinoma at stages I-II: The patients underwent sentinel node biopsy and posterior neck dissection
  Interventions: Procedure: Sentinel node biopsy guided by magnetic probe

INTERVENTIONS:
Procedure: Sentinel node biopsy guided by magnetic probe — Sentinel nodes exeresis guided by magnetic probe after injection submucosally and peritumorally of super-para-magnetic contrast. Standard neck dissection (levels I-II) were carry out after sentinel node biopsy

SUMMARY:
Sentinel node biopsy has been shown to be a viable alternative to elective neck dissection in the early stages of squamous cell oral carcinoma. The aim of this study was to describe the magnetic localization of sentinel nodes (SN) after peritumoral injection of superparamagnetic iron oxide (SPIO) for treating this type of tumor and to analyze the technique's diagnostic performance in 23 patients. The technique located SNs (with minimal complication) in 95.6 % (22/23) of the patients. Three relapses occurred, one in a patient who had shown negative in magnetic SN location and elective neck dissection. The diagnostic performance of magnetic localization achieved a sensitivity and negative predictive value of 0.80 y 0.94, respectively. Magnetic localization of SNs has been shown to be a reproducible technique that may offer a viable alternative to the conventional technique.

ELIGIBILITY:
Inclusion Criteria:

* Oral squamous cell carcinoma T1-T2, cN0.
* Absence of alterations to iron metabolism.

Exclusion Criteria:

* Previous neck surgery.
* Treatment with iron chelators.
* Pregnant

Ages: 29 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited consecutively when diagnosed with oral squamous cell carcinoma at clinical stages I-II by biopsy and magnetic resonance. All patients were intervened by the same surgeon at the Department of Maxillofacial Surgery at Donostia University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of SNB was analyzed in terms of sensitivity (S), specificity (Sp), negative and positive predictive value (NPV and PPV). | Six years

CONTACTS AND LOCATIONS:
Locations (1):
- Josué Hernando Vázquez, Donostia / San Sebastian, Guipuzkoa, Spain